CLINICAL TRIAL: NCT00632476
Title: In-Utero Smoke, Vitamin C, and Newborn Lung Function
Brief Title: Evaluating the Effects of Supplemental Vitamin C on Infant Lung Function in Pregnant Smoking Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); National Institute of Environmental Health Sciences (NIEHS) (NIH)
Responsible Party: Principal Investigator, Cynthia McEvoy, Associate Professor of Pediatrics, National Heart, Lung, and Blood Institute (NHLBI)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 546; K23HL080231 (NIH); K23HL080231-01A1 (NIH)
Record Dates: First submitted 2008-03-05; First posted 2008-03-10 (Estimated); Last update posted 2013-09-04 (Estimated); Status verified 2013-08

CONDITIONS: Pregnancy; Smoking
Keywords: Smoking During Pregnancy; Vitamin C; Newborn Lung Function; Ascorbic Acid
MeSH Terms: conditions — Smoking | interventions — Sugars; Ascorbic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- A (Placebo Comparator): Participants will receive a placebo capsule throughout pregnancy.
  Interventions: Other: Placebo
- B (Active Comparator): Participants will receive a vitamin C capsule throughout pregnancy.
  Interventions: Dietary Supplement: Vitamin C
- C (No Intervention): A group of non-smoking pregnant women will not receive placebo or vitamin C.

INTERVENTIONS:
Other: Placebo — Placebo capsule once a day
  Other Names: Sugar pill
  Arms: A
Dietary Supplement: Vitamin C — A 500-mg vitamin C capsule once a day
  Other Names: Ascorbic acid
  Arms: B

SUMMARY:
Women who smoke during their pregnancy place their unborn child at an increased risk of health problems, including decreased lung function and possible lung diseases later in life. Preliminary animal research suggests that if vitamin C is taken during pregnancy, nicotine's harmful effects on the unborn baby's developing lungs may be blocked. This study will determine the effect that vitamin C has on the lung development and function of babies born to women who smoke during pregnancy.

DETAILED DESCRIPTION:
Approximately 12% of women smoke during pregnancy, and at least 500,000 babies are born each year having been exposed to nicotine. These infants have poor lung function at birth and have an increased risk of developing lung diseases, including bronchitis, pneumonia, and asthma. Researchers believe that nicotine may interact with nicotinic receptors in the unborn child's developing lungs and cause altered growth and decreased lung function. Preliminary animal research studies suggest that some of the harmful effects of nicotine may be blocked by vitamin C, an antioxidant that may protect against cellular damage caused by nicotine and other pollutants. The purpose of this study is to evaluate the effectiveness of vitamin C at blocking the harmful effects of nicotine exposure on lung development and function in children born to women who smoke during pregnancy.

This study will enroll pregnant women who smoke, as well as a control group of pregnant women who do not smoke. At a baseline study visit, all participants will complete smoking history questionnaires. For 2 weeks, all participants who smoke will receive placebo capsules once a day. They will then be randomly assigned to receive either vitamin C capsules or placebo capsules, both of which will be taken once a day, in addition to a prenatal vitamin, for the duration of their pregnancy. Study visits, occurring once a month throughout the pregnancy, will include a medical and smoking history review and urine collection. An ultrasound exam will be performed once during the pregnancy to determine the exact size and age of the baby, and blood collection will occur at baseline and once or twice more during the pregnancy. Study researchers will review participants' medical records and will call participants three times during their pregnancy to review their food intake. At the time of delivery, amniotic fluid samples will be collected. When babies are 48 hours old, baby lung function testing will occur, and when babies are 3 and 9 months of age, researchers will call participants to collect breathing information on the babies. When babies are 12 months old, participants will attend a study visit that will include urine collection from the babies and a review of baby breathing difficulties, medication changes, and environmental smoking exposure.

ELIGIBILITY:
Inclusion Criteria:

* Randomly assigned to a study intervention at less than 22 weeks of gestation
* History of smoking
* Singleton gestation pregnancy
* Smoking cessation intervention offered but declined

Exclusion Criteria:

* Multiple gestation pregnancy
* Documented major fetal congenital anomalies
* History of kidney stones
* Insulin dependent diabetes
* Current participation in other research projects that may interfere with this study
* Continuous use of high dose vitamin C since last menstrual period (LMP) or initial ascorbic acid level greater than 100 micromoles/liter

Min Age: 15 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 282 (Actual)
Dates: Start 2007-03; Primary Completion 2011-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Pulmonary function testing (including respiratory compliance and the ratio of time to peak tidal expiratory flow to total expiratory time) | Measured within 48 hours after delivery

SECONDARY OUTCOMES:
Pulmonary function testing (including respiratory compliance and the ratio of time to peak tidal expiratory flow to total expiratory time)and respiratory history including wheezing through 12 months of age. | Measured at 12 months of age

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia T. McEvoy, MD, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health & Science University, Portland, Oregon, United States

REFERENCES:
- [Derived] Shorey-Kendrick LE, McEvoy CT, Ferguson B, Burchard J, Park BS, Gao L, Vuylsteke BH, Milner KF, Morris CD, Spindel ER. Vitamin C Prevents Offspring DNA Methylation Changes Associated with Maternal Smoking in Pregnancy. Am J Respir Crit Care Med. 2017 Sep 15;196(6):745-755. doi: 10.1164/rccm.201610-2141OC. PMID 28422514
- [Derived] McEvoy CT, Schilling D, Clay N, Jackson K, Go MD, Spitale P, Bunten C, Leiva M, Gonzales D, Hollister-Smith J, Durand M, Frei B, Buist AS, Peters D, Morris CD, Spindel ER. Vitamin C supplementation for pregnant smoking women and pulmonary function in their newborn infants: a randomized clinical trial. JAMA. 2014 May;311(20):2074-82. doi: 10.1001/jama.2014.5217. PMID 24838476
- [Derived] Didenco S, Gillingham MB, Go MD, Leonard SW, Traber MG, McEvoy CT. Increased vitamin E intake is associated with higher alpha-tocopherol concentration in the maternal circulation but higher alpha-carboxyethyl hydroxychroman concentration in the fetal circulation. Am J Clin Nutr. 2011 Feb;93(2):368-73. doi: 10.3945/ajcn.110.008367. Epub 2010 Dec 15. PMID 21159788